CLINICAL TRIAL: NCT06506786
Title: Microbiomes of Garden-fresh vs Store-bought Produce and Variation in Their Effects on the Human Gut Microbiome
Brief Title: Garden-fresh Foods and Gut Microbiomes
Acronym: GFF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oregon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2023-67017-39054
Record Dates: First submitted 2024-05-24; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Gut Microbiome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Garden First (Experimental): Participants assigned to this study arm undergo the Garden-fresh Produce intervention during the first period and the Supermarket Produce intervention during the second period.
  Interventions: Other: Garden-fresh Produce; Other: Supermarket Produce
- Supermarket First (Experimental): Participants assigned to this study arm undergo the Supermarket Produce intervention during the first period and the Garden-fresh Produce intervention during the second period.
  Interventions: Other: Garden-fresh Produce; Other: Supermarket Produce

INTERVENTIONS:
Other: Garden-fresh Produce — Participants are asked to consume the USDA-recommended amounts of fruits and vegetables harvested from their gardens.
Other: Supermarket Produce — Participants are asked to consume the USDA-recommended amounts of fruits and vegetables purchased from a supermarket.

SUMMARY:
The purpose of this research is to explore what types of microbes are present on garden-fresh versus store-bought fruits and vegetables, as well as how they might affect the human gut microbiome.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Body mass index (BMI) greater than or equal to 35 or less than or equal to 18.
* Age under 18 or over 45.
* Female who is pregnant or lactating.
* Irregular bowel movements and/or stool consistency.
* Plans to travel, move residences, or other major life change during the study period (August-October 2023).
* Unable to speak, read, and write English.
* Use of any of the following drugs within the last 6 months:
* systemic antibiotics, antifungals, antivirals or antiparasitics (intravenous, intramuscular, or oral);
* oral, intravenous, intramuscular, nasal or inhaled corticosteroids;
* cytokines;
* methotrexate or immunosuppressive cytotoxic agents;
* large doses of commercial probiotics consumed (greater than or equal to 108 cfu or organisms per day) - includes tablets, capsules, lozenges, chewing gum or powders in which probiotic is a primary component. Ordinary dietary components such as fermented beverages/milks, yogurts, foods do not apply.
* Acute disease at the time of enrollment (defer sampling until subject recovers). Acute disease is defined as the presence of a moderate or severe illness with or without fever.
* History of cancer except for squamous or basal cell carcinomas of the skin that have been medically managed by local excision.
* Unstable dietary history as defined by major changes in diet during the previous month, where the subject has eliminated or significantly increased a major food group in the diet.
* Recent history of chronic alcohol consumption defined as more than five 1.5-ounce servings of 80 proof distilled spirits, five 12-ounce servings of beer or five 5-ounce servings of wine per day.
* Any confirmed or suspected condition/state of immunosuppression or immunodeficiency (primary or acquired) including HIV infection.
* Major surgery of the GI tract, with the exception of cholecystectomy and appendectomy, in the past five years. Any major bowel resection at any time.
* History of active uncontrolled gastrointestinal disorders or diseases including:
* inflammatory bowel disease (IBD) including ulcerative colitis (mild-moderate-severe), Crohn's disease (mild-moderate-severe), or indeterminate colitis;
* irritable bowel syndrome (IBS) (moderate-severe);
* persistent, infectious gastroenteritis, colitis or gastritis, persistent or chronic diarrhea of unknown etiology, Clostridium difficile infection (recurrent) or Helicobacter pylori infection (untreated);
* chronic constipation.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference in fecal bacterial abundance, as characterized by qPCR with "universal" bacterial primers | Baseline, 1 week, 3 weeks
  ANOVA statistical test of bacterial gene copies (a proxy for absolute abundance) used to compare whether Garden-Fresh Produce and Supermarket Produce interventions differentially affect fecal bacterial abundance.
Difference in fecal microbial diversity, as characterized by shotgun metagenomics. | Baseline, 1 week, 3 weeks
  ANOVA statistical test of Shannon index used to compare whether Garden-Fresh Produce and Supermarket Produce interventions differentially affect fecal microbial diversity.
Difference in fecal microbial composition, as characterized by shotgun metagenomics. | Baseline, 1 week, 3 weeks
  PERMANOVA statistical test used to compare whether Garden-Fresh Produce and Supermarket Produce interventions differentially affect fecal microbial composition.
Presence of differentially abundant microbial taxa, as characterized by shotgun metagenomics. | Baseline, 1 week, 3 weeks
  Negative binomial GLM statistical test used to identify microbial taxa associated with either Garden-Fresh Produce or Supermarket Produce intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Gwynne Mhuireach, PhD, Principal Investigator — University of Oregon
Locations (1):
- Institute for Health in the Built Environment, University of Oregon, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: No